CLINICAL TRIAL: NCT01594554
Title: A 5-year Observational Follow-up Study to Describe Treatment Patterns and Outcomes in Real World Clinical Practice for Patients of Newly Confirmed HCV Infection in China (2012-2016)
Brief Title: A 5-year Observational Follow-up Study to Describe Treatment Patterns in Real World of HCV Patients in China.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Lai Wei, Director of Peking University Hepatology Institute at Peking University People's Hospital, Peking University People's Hospital
Other Study IDs: AI452018 ST; CCgenos Follow-up phase (Other: EC of Peking University People's Hospital)
Record Dates: First submitted 2012-04-04; First posted 2012-05-09 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Hepatitis C
Keywords: HCV viral genotypes; host genotypes; IL28B; Outcome; Follow-Up; ITPA; RNA; China
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with HCV RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV Patients: A sample of 600 Han ethnic Chinese male or female who are ≥ 18 years old enrolled and completed in the study of AI452-009 (i.e., CCgenos cross sectional phase, ClinicalTrials.gov Identifier: NCT01293279).

SUMMARY:
A 5-year study to observe and describe long-term patient management and treatment patterns with associated outcomes of patients who previously enrolled in Protocol AI452009 (i.e., the CCgenos cross sectional phase, ClinicalTrials.gov Identifier: NCT01293279) and had their genotype characterized at diagnosis of HCV infection in a real world clinical practice in China.

DETAILED DESCRIPTION:
A sample of 600 Han ethnic Chinese male or female who are ≥ 18 years old enrolled and completed in the study of AI452-009 (i.e., CCgenos cross sectional phase, ClinicalTrials.gov Identifier: NCT01293279). In the AI452-009 study, all patients had a recent confirmation of anti-HCV-antibody positive and HCV RNA positive but antiviral treatment naive from 28 university affiliated hospital in China. The primary objective of this study (AI452-018, CCgenos follow up phase, ClinicalTrials.gov Identifier: NCT01293279) is to observe and describe long-term patient management and treatment patterns with associated outcomes of patients who previously enrolled in Protocol AI452009 (i.e., the CCgenos cross sectional phase, ClinicalTrials.gov Identifier: NCT01293279) and had their genotype characterized at diagnosis of HCV infection in a real world clinical practice in China.

ELIGIBILITY:
Inclusion Criteria:

* None. Patients from AI452-009 study who accepted ICF to be follow up

Exclusion Criteria:

* < 18 years old not Han ethnic Not be willing to be followed up to 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
HCV RNA level | 5 years
  • HCV RNA level when on HCV treatments

SECONDARY OUTCOMES:
Subjects ratio of cirrhosis, HCC and death | 5 years
  • Evaluation of HCV disease progression (cirrhosis, HCC, death) over time regardless treatment options
Viral genotypes of subjects | 5 years
  Evaluation of impacts of risk factors, such as viral genotypes on disease progression overtime
Host genotypes of subjects | 5 years
  Evaluation of impacts of risk factors, such as host genotypes on disease progression overtime
Diabetes status of subjects | 5 years
  Evaluation of impacts of risk factors, such as diabetes status on disease progression overtime

CONTACTS AND LOCATIONS:
Overall Officials: Hong Li, Ph.D, Study Director — Bristol-Myers Squibb
Locations (1):
- Wei Lai, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Huang R, Shang J, Chen H, Li J, Xie Q, Feng J, Wei L, Rao H. Sustained virologic response improved the long-term health-related quality of life in patients with chronic hepatitis C: a prospective national study in China. BMC Infect Dis. 2024 Jan 10;24(1):72. doi: 10.1186/s12879-023-08940-3. PMID 38200419
- [Derived] Wu N, Rao HY, Yang WB, Gao ZL, Yang RF, Fei R, Gao YH, Jin Q, Wei L. Impact of hepatitis C virus genotype 3 on liver disease progression in a Chinese national cohort. Chin Med J (Engl). 2020 Feb 5;133(3):253-261. doi: 10.1097/CM9.0000000000000629. PMID 31934936
- [Derived] Rao H, Xie Q, Shang J, Gao Z, Chen H, Sun Y, Jiang J, Niu J, Zhang L, Wang L, Zhao L, Li J, Yang R, Zhu S, Li R, Wei L. Real-world clinical outcomes among individuals with chronic HCV infection in China: CCgenos study. Antivir Ther. 2019;24(7):473-483. doi: 10.3851/IMP3334. PMID 31566575